CLINICAL TRIAL: NCT03788798
Title: An Integrated Model of Intelligent Medical Service for Total Joint Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 104-8598B
Record Dates: First submitted 2018-12-13; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-03

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical pathway (No Intervention): A standard clinical pathway for TKA has been compulsively implemented for medical cost containment and quality assurance to meet with the Taiwan Diagnosis-Related Groups (TW-DRGs) payment system since 1997. The clinical pathway for TKA undertakes with preadmissions, anesthetic, surgery, and physiotherapy assessment. Medical, nursing, and physiotherapy assessment were put down for each postadmission day. The time from admission to surgery, the use of intravenous antibiotics injection and intravenous fluid were all assessed. Discharge criteria were active knee flexion to 90 degrees, having the ability to walk with aids and clean wound condition with any infection sign. The pathway was initially set for a 6-day postoperative length of stay.
- Patient Infotainment Terminal (Experimental): Patients who have additional access to an integrated infotainment system and are cared by a standard clinical pathway. The patient infotainment system is a quasi-interactive computer program connected to a server that pushes messages and educational programs ordered from the caring physicians or on-demand by the patients. The server has parallel data exchange gateways to the Hospital Information System (HIS), Picture Archiving Communication System (PACS), and can record the patients' responses to surveys and questionnaires.
  Interventions: Device: Patient infotainment system

INTERVENTIONS:
Device: Patient infotainment system — The patient infotainment system is a quasi-interactive computer program connected to a server that pushes messages and educational programs ordered from the caring physicians or on-demand by the patients. The server has parallel data exchange gateways to the Hospital Information System (HIS), Picture Archiving Communication System (PACS), and can record the patients' responses to surveys and questionnaires.
  Arms: Patient Infotainment Terminal

SUMMARY:
With the aging population, the needs for total joint replacement are increasing. A successful recovery after joint replacement surgery depends on timely and active physical therapy in the early postoperative period. To accomplish it, an integrated care model based on clinical pathway has been implemented to secure the medical quality and patient safety. Recently, the emerging technology of electronic medical record and medical informatics have made challenges to the traditional health care models such as the clinical pathway. As a matter of fact, the integration of informatics technology also provides an opportunity to modernize the clinical pathway and make it smarter. By bridging the HIS system and the medical cloud of a virtual platform of interactive clinical pathway, the quality of care and patient safety can be better secured and the performance can be stored for analysis.

The project " The effects of intelligent clinical pathway for total joint replacement" is a subproject of the integrated project " An integrated model of intelligent medical service for total joint replacement". It will be carried out in a facility built with intelligent environment (Kaohsiung CGMH) and the data will be stored and computed in the medical care cloud and specialist system server. Collaborating with subproject 2 and 4 (smart wearing device) and subproject 3 (total nursing care), this project is intended to set the milestones for the postoperative recovery after total joint replacement. Supplemented with the specialist system and interactive programs, it will be implemented in total joint replacement patients as an vehicle for perioperative assessment, follow-up, monitoring, and instruction. The big data of the objective analytic results and feedback from the patients will be the important reference for medical and health promotion.

DETAILED DESCRIPTION:
With the aging population, the needs for total joint replacement are increasing. On the basis of 2000-to-2014 data from National Inpatient Sample (NIS), primary total knee arthroplasty (TKA) is projected to grow by 85% to 1.26 million procedures in the United States by 2030. In a 2012 report of Orthopaedic Industry, and the global sales of joint replacement products exceeded $49.3 billion, with knees taking about half of them. The high financial burden of joint replacement surgery on health care system highlights the importance of cost containment without compromising the quality of patient care.

Clinical pathways for total joint arthroplasty can reduce care variability and improve the quality of care. Taiwan's Bureau of National Health Insurance (BNHI) has initiated a prospective payment system for TKA under diagnosis-related group (DRG) since 1997. It was found the length of hospital stay, and the medical expenditure could be reduced because standard clinical pathways were implemented in most hospitals. However, to optimize the results and meet with patients' expectation are more challenging currently than before because the length of hospitalization is markedly reduced and the standard care processes are accelerated. The accelerated programs for total joint arthroplasty are revolutionizing the standard clinical pathways. Patients can even be discharged from the hospital within one day after the surgery. While a successful joint replacement surgery depends on well-practiced clinical pathways delivered in a timely manner, patient's medical literacy should also have a significant impact for his or her recovery. Unfortunately, patients may acquire incorrect information from the internet or have unrealistic expectations before or during the hospitalization that may compromise the decision making and clinical results.

Recently, the emerging technologies of the electronic medical record and medical informatics have made challenges to the traditional healthcare models such as the clinical pathways. The integration of informatics technology also provides an opportunity to modernize the clinical pathways. But the effect of an interactive infotainment system on TKA is unknown. The purpose of this study was to analyze whether the implementation of an interactive infotainment system into a standard clinical pathway of TKA could influence the hospital course and the medical quality in an arthroplasty specialty ward.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the hospital, scheduled for total joint replacement surgery
* Sign informed consent form

Exclusion Criteria:

* In-patient, not scheduled for total joint replacement surgery
* Any psychological condition or other condition that may influence the study result

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Length of stay | up to 10 days
  in hospital stay (days)
30-day return to emergency room | within 30 days after discharge
  Patients who will return to the emergency room within 30 days after discharge
30-day readmission after discharge | within 30 days after discharge
  Patients who will readmit within 30 days after discharge
90-day return to emergency room | within 90 days after discharge
  Patients who will return to the emergency room within 90 days after discharge
90-day readmission after discharge | within 90 days after discharge
  Patients who will readmit within 90 days after discharge

SECONDARY OUTCOMES:
medical expenditure | up to 10 days
  The total medical cost in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mel S Lee, MD,PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No